CLINICAL TRIAL: NCT03403556
Title: A Randomized, Multicenter, Open, Parallel, Phase 4 Study to Compare the Efficacy and Safety Between High-intensity Rosuvastatin and Moderate-intensity Rosuvastatin/Ezetimibe in High ASCVD Risk Patients With Type 2 diabEtes (CREATE Study)
Brief Title: High-intensity Rosuvastatin vs. Moderate-intensity Rosuvastatin/Ezetimibe in High Atherosclerotic Cardiovascular Disease Risk Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREATE
Record Dates: First submitted 2017-12-11; First posted 2018-01-18 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Atherosclerotic Cardiovascular Disease; Type 2 Diabetes
Keywords: High ASCVD risk patients with type 2 diabetes
MeSH Terms: conditions — Atherosclerosis; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvamibe ® Tab. (Experimental): Rosuvastatin 10mg/Ezetimibe10mg
  Interventions: Drug: Rosuvamibe
- Monorova ® Tab. (Active Comparator): Rosuvastatin 20mg
  Interventions: Drug: Monorova

INTERVENTIONS:
Drug: Rosuvamibe — Rosuvastatin 10mg/Ezetimibe10mg qd for 24 weeks
  Arms: Rosuvamibe ® Tab.
Drug: Monorova — Rosuvastatin 20mg qd for 24 weeks
  Arms: Monorova ® Tab.

SUMMARY:
To assess the efficacy and safety of moderate-intensity rosuvastatin/ezetimibe compared to high-intensity rosuvastatin in high atherosclerotic cardiovascular disease risk patients with type 2 diabetes

DETAILED DESCRIPTION:
This study is to assess the efficacy and safety of Rosuvamibe® (rosuvastatin 10mg/ezetimibe 10mg) vs. rosuvastatin 20mg treated for 24 weeks in atherosclerotic cardiovascular disease risk (≥ 7.5%) patients with type 2 diabetes

ELIGIBILITY:
* ≥ 40 and < 75 years of age at the time of informed consent
* Estimated 10-year ASCVD (atherosclerotic cardiovascular disease) risk ≥ 7.5% with type 2 diabetes according to the American Diabetes Association criteria in screening
* HbA1c ≥ 6% and < 10% in screening
* Body mass index (BMI) ≤ 35kg/m2 in screening
* Female of childbearing with a negative pregnancy test who must agree to use contraception (including those not medically pregnant) during the study period
* Written consent after being informed of the purpose and contents of the clinical trial and the characteristics and risks of IPs

Exclusion Criteria:

* Type 1 diabetes
* Chronic hepatitis B or chronic hepatitis C, severe hepatic dysfunction (AST, ALT, ALP or CPK ≥ 3 x ULN) in screening
* Heavy drinking > 210g per week in screening
* Estimated GFR < 30mL/min/1.73m2 using the CKD-EPI formula in screening
* Undergoing renal replacement therapy (hemodialysis or peritoneal dialysis) in screening
* Having used other statin (HMG-CoA converting enzyme inhibitors) than Rosuvastatin or fibrate drugs in the last 3 months before screening
* Taking any medication (ex. Fenofibrate, Omega 3 fatty acid, etc.) that may affect LDL

  * Can be enrolled after 4 week-washout
* Having used thiazolidinedione drugs in the last 3 months before screening
* Taking cyclosporine concomitantly
* Positive HIV test in screening
* Pregnant, breastfeeding, or childbearing women who are not likely to use the appropriate contraceptive methods as judged by investigator
* Subjects with a medical history of myopathy and rhabdomyolysis due to use of statin
* Hypersensitive to statin and ezetimibe
* Having endocrine or metabolic disease known to affect serum lipids or lipoproteins

  * Uncontrolled diabetes (HbA1c ≥ 10%)
  * Uncontrolled thyroid dysfunction (TSH ≥ 3 x ULN)
* Subjects with a medical history of acute arterial diseases such as unstable angina, myocardial infarction, transient ischemic attack, cerebrovascular disease, coronary artery bypass graft or percutaneous coronary intervention in the last 6 months before screening
* Subjects with a surgical history of gastrointestine or drug absorption disorders due to gastrointestinal disorders
* Insulin-treated
* Taking other IPs in the last 30 days before screening
* Subjects who cannot discontinue contraindications that may affect the treatment of all types of diabetes and/or hypercholesterolemia during the study period
* Subjects with a significant or unstable medical or psychological condition that is judged by investigator to be detrimental to safety or to successful participation in the trial
* Other conditions than the above who is deemed to be ineligible to participate in the trial by investigator

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-03-27 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Mean percent change from baseline to week 24 in low-density lipoprotein cholesterol (LDL-C) | Up to 24 weeks

SECONDARY OUTCOMES:
Proportion of subjects achieving < 7.5% 10-year ASCVD risk without withdrawn due to adverse events | Up to 24 weeks
Mean change from baseline to week 12 and to week 24 in 10-year ASCVD risk | Up to 12 weeks, Up to 24 weeks
Proportion of subjects achieving the comprehensive lipid target (LDL-C < 70mg/dL, Non-HDL-C < 100mg/dL, and Apolipoprotein B < 80mg/dL) without withdrawn due to adverse events | Up to 24 weeks
Mean change from baseline to week 24 in calculated LDL cholesterol(mg/dL), HDL cholesterol(mg/dL), Triglyceride(mg/dL), non-HDL cholesterol(mg/dL), Apolipoprotein B(mg/dL), Apolipoprotein A1(mg/dL) | Up to 24 weeks
Mean change from baseline to week 24 in Hepatic Steatosis Index (HSI) | Up to 24 weeks
  hepatic steatosis index (HSI)= 8x(ALT/AST ratio)+BMI (+2, if female; +2, if diabetes mellitus)
Mean change from baseline to week 24 in Fatty Liver Index (FLI) | Up to 24 weeks
  FLI scores will be calculated based on triglycerides, BMI, r-GT and Waist circumference. BMI(kg/m^2) will be calculated based on height(m) and weight(kg).
Mean change from baseline to week 24 in non-alcoholic fatty liver disease liver fat score (NAFLD-LFS) | Up to 24 weeks
Mean change from baseline to week 24 in HbA1c | Up to 24 weeks
Mean change from baseline to week 24 in fasting plasma glucose (FPG) | Up to 24 weeks
Mean change from baseline to week 24 in sCD36 | Up to 24 weeks
Mean change from baseline to week 24 in HOMA-IR | Up to 24 weeks
Mean change from baseline to week 24 in HOMA-B | Up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - The Catholic University of Korea, St. Vincent's Hospital, Gyeonggi-do
  - Korea University Anam Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No